CLINICAL TRIAL: NCT06932991
Title: Cognitive Stimulation Therapy vs. Reality Orientation & Reminiscence Therapy: Effects on Cognitive and Functional Domains in Dementia - Retrospective Study
Brief Title: Cognitive Stimulation Therapy - Effects on Cognitive and Functional Domains in Dementia - A Retrospective Data Review
Acronym: CST
Status: Completed | Type: Observational
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Frank Lai, Assistant Professor, Northumbria University
Other Study IDs: CST - Retrospective Datareview
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-04

CONDITIONS: Dementia
Keywords: older adults; dementia
MeSH Terms: conditions — Dementia | interventions — Cognitive Remediation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cognitive Stimulation Therapy: Therapy in the CST arm focused on improving participants' attention span, memory and problem-solving skills using paper and pen, table games or computer programs.
  Interventions: Behavioral: Cognitive Remediation
- RO&RM arm: with the use of orientation boards, calendars, clocks, verbal reminders, and different environmental cues to reduce participants' confusion, disorientation and behavioral problems.
  Interventions: Behavioral: Cognitive Remediation

INTERVENTIONS:
Behavioral: Cognitive Remediation — cognitive remediation

SUMMARY:
This retrospective, single-blind, parallel group study investigates the efficacy of Cognitive Stimulation Therapy (CST) compared to Reality Orientation and Reminiscence Therapy (RO&RM) in enhancing cognitive and functional domains in older adults with mild to moderate dementia.

DETAILED DESCRIPTION:
Through data review, this retrospective, single-blind, parallel group study investigates the efficacy of Cognitive Stimulation Therapy (CST) compared to Reality Orientation and Reminiscence Therapy (RO&RM) in enhancing cognitive and functional domains in older adults with mild to moderate dementia.

ELIGIBILITY:
Inclusion Criteria:

* participants had to be 65 years old or above, live in Hong Kong and had a diagnosis for dementia in medical history

Exclusion Criteria:

* any major neurological illness other than dementia, any psychiatric disorder or a known history of substance abuse.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older people who are residence in a 24/7 care home
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Kendrick Cognitive Test for the Elderly (KCTE). | Baseline line and six-month
  Participants' attention and episodic memory were quantified using the Kendrick Cognitive Test for the Elderly (KCTE).

SECONDARY OUTCOMES:
The Chinese Disability Assessment for Dementia (CDAD) | Baseline and 6-month after the start of the program
  for assessing executive function in older adults with dementia. Its focus on initiating, planning, and executing activities provides a practical and ecologically valid measure of executive dysfunction, aligning closely with the real-world challenges faced by older Chinese people with dementia.

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria University, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spector A, Thorgrimsen L, Woods B, Royan L, Davies S, Butterworth M, Orrell M. Efficacy of an evidence-based cognitive stimulation therapy programme for people with dementia: randomised controlled trial. Br J Psychiatry. 2003 Sep;183:248-54. doi: 10.1192/bjp.183.3.248. PMID 12948999
- [Background] Mok CC, Siu AM, Chan WC, Yeung KM, Pan PC, Li SW. Functional disabilities profile of chinese elderly people with Alzheimer's disease - a validation study on the chinese version of the disability assessment for dementia. Dement Geriatr Cogn Disord. 2005;20(2-3):112-9. doi: 10.1159/000086612. Epub 2005 Jun 30. PMID 15990425